CLINICAL TRIAL: NCT03225339
Title: A Randomised Controlled Trial Assessing the Impact of Low Calorie Diet and Activity on Body Weight and Glycaemia in Diabetes
Brief Title: Diabetes Intervention Accentuating Diet and Enhancing Metabolism
Acronym: DIADEM-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Cornell Medical College in Qatar (Other)
Collaborators: Hamad Medical Corporation (Industry); Weill Medical College of Cornell University (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-00071
Record Dates: First submitted 2017-06-12; First posted 2017-07-21 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All analyses conducted will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Intervention (Experimental): The intervention includes the use of Low Energy Diet replacement products in combination with physical activity, followed by gradual introduction of food, and increasing physical activity. Behavioural support for the lifestyle intervention will also be provided.
  Interventions: Dietary Supplement: Low Energy Diet
- Usual Care (No Intervention): This will be based on current clinical practice aiming to reduce diabetes symptoms and complications, and general recommendations on diet and physical activity.

INTERVENTIONS:
Dietary Supplement: Low Energy Diet — Low Energy Diet
  Arms: Lifestyle Intervention

SUMMARY:
Diabetes is one of the greatest challenges faced by healthcare services worldwide. It is associated with serious complications such as heart attacks, stroke, and peripheral artery disease as well as kidney disease, eye disease, and nerve dysfunction. Data from weight loss with bariatric surgery suggest that with the appropriate intervention, it should be possible to reverse diabetes and that the earlier the intervention occurs, the greater the chances of placing diabetes into remission. There is now a need to translate this knowledge into the medical care of younger patients with early diabetes who are overweight/obese. The aim of this study is to see if younger adult patients with overweight/obesity and type 2 diabetes who are participants in a programme incorporating a low energy diet and physical activity (lifestyle) will lower their weight, cardiovascular risk and improve their glycaemic control as compared to the usual care.

DETAILED DESCRIPTION:
The aim of the proposed study is to conduct a pragmatic randomised controlled clinical trial randomising young adult patients with obesity and type 2 diabetes to an intervention incorporating a low calorie diet and physical activity or usual care. The investigators hypothesise that patients in the low calorie intervention arm will have greater weight reduction leading to significant improvement in glycaemic control and cardiovascular risk. The primary outcome will be weight loss. The low calorie diet intervention arm is designed to achieve and maintain significant weight loss through decreased calorie intake, increased physical activity, and behaviour change. Usual care will include routine advice about diet and physical activity. Secondary outcomes include diabetes control, body composition, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (based on ADA diagnostic criteria) ;
* Diabetes of ≤ 3-year duration;
* BMI >27.0 kg/m² (based on WHO cut-points for ethnicity 119);
* Men and women;
* Age 18-50 years;
* Originating from the Middle East and North Africa region and resident in Qatar;
* Able to commit to the study duration;
* Able to give informed consent and willing to participate in the study.

Exclusion Criteria:

* Type 1 diabetes mellitus based on clinical history;
* Cardiovascular event in the previous 6 months;
* Chronic kidney disease stage 3b or greater (eGFR <30 mL/min/1.73m²);
* Currently pregnant, lactating, or planning pregnancy within the study period;
* Any condition precipitating fluid overload such as heart failure (NYHA class > I) and liver cirrhosis;
* Significant previously diagnosed psychiatric disorder (e.g. schizophrenia, post-traumatic stress disorder, obsessive-compulsive disorder);
* Uncontrolled depression (based on hospital anxiety and depression scale);
* Uncontrolled epilepsy;
* Known lactose intolerance;
* Severe arthritis preventing walking;
* Active gout;
* Active gallstone disease or known asymptomatic gallstones.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2017-07-16 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Weight loss | 12 months
  Weight change (weight in kilograms)

SECONDARY OUTCOMES:
Glycaemic control | 12 months
  HbA1c measured biochemically (percentage units)
Patient reported outcomes | 12 months
  Euro-QoL-5D

OTHER OUTCOMES:
Insulin sensitivity/resistance | 12 months
  Fasting Insulin and Glucose levels will be combined to calculate:
  Homeostatic model assessment (HOMA-IR)
Body Mass Index | 12 months
  Weight and height measures will be used to calculate body mass index: Weight(kg)/(height[m])2
Waist Circumference | 12 months
  Waist Circumference measured in cm

CONTACTS AND LOCATIONS:
Overall Officials: Shahrad Taheri, MB BS PhD, Principal Investigator — Weill Cornell Medicine - Qatar
Locations (2):
- Qatar (2):
  - Primary Healthcare Corporation, Doha
  - Hamad Medical Corporation, Doha

IPD SHARING:
Plan to Share IPD: Yes
Data will be available from the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2022-2024
Access Criteria: Access requests to be made to the Principal Investigator.

REFERENCES:
- [Background] Taheri S, Chagoury O, Zaghloul H, Elhadad S, Ahmed SH, Omar O, Payra S, Ahmed S, El Khatib N, Amona RA, El Nahas K, Bolton M, Chaar H, Suleiman N, Jayyousi A, Zirie M, Janahi I, Elhag W, Alnaama A, Zainel A, Hassan D, Cable T, Charlson M, Wells M, Al-Hamaq A, Al-Abdulla S, Abou-Samra AB. Diabetes Intervention Accentuating Diet and Enhancing Metabolism (DIADEM-I): a randomised controlled trial to examine the impact of an intensive lifestyle intervention consisting of a low-energy diet and physical activity on body weight and metabolism in early type 2 diabetes mellitus: study protocol for a randomized controlled trial. Trials. 2018 May 21;19(1):284. doi: 10.1186/s13063-018-2660-1. PMID 29784059
- [Result] Taheri S, Zaghloul H, Chagoury O, Elhadad S, Ahmed SH, El Khatib N, Amona RA, El Nahas K, Suleiman N, Alnaama A, Al-Hamaq A, Charlson M, Wells MT, Al-Abdulla S, Abou-Samra AB. Effect of intensive lifestyle intervention on bodyweight and glycaemia in early type 2 diabetes (DIADEM-I): an open-label, parallel-group, randomised controlled trial. Lancet Diabetes Endocrinol. 2020 Jun;8(6):477-489. doi: 10.1016/S2213-8587(20)30117-0. PMID 32445735
- [Derived] Zaghloul H, Chagoury O, Elhadad S, Hayder Ahmed S, Suleiman N, Al Naama A, El Nahas K, Al Hamaq A, Charlson M, Wells MT, Al Abdulla S, Abou-Samra AB, Taheri S. Clinical and metabolic characteristics of the Diabetes Intervention Accentuating Diet and Enhancing Metabolism (DIADEM-I) randomised clinical trial cohort. BMJ Open. 2020 Dec 7;10(12):e041386. doi: 10.1136/bmjopen-2020-041386. PMID 33293319